CLINICAL TRIAL: NCT00654914
Title: A National, Multicentre, Open Label, Flexible Dose, Twelve Week Treatment to Assess the Efficacy and Safety of 5mg, 10mg and 20mg Bay 38-9456, a Phosphodiesterase Type V Inhibitor, in the Treatment of Male Patients With Erectile Dysfunction
Brief Title: A Study to Assess the Efficacy and Safety of Vardenafil in the Treatment of Male Patients With Erectile Dysfunction
Acronym: VIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10781
Record Dates: First submitted 2008-04-04; First posted 2008-04-09 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Erectile Dysfunction
Keywords: Sexual Dysfunction
MeSH Terms: conditions — Erectile Dysfunction; Sexual Dysfunction, Physiological | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Levitra (Vardenafil, BAY38-9456)

INTERVENTIONS:
Drug: Levitra (Vardenafil, BAY38-9456) — 10 mg per dose of vardenafil for the first four weeks. A further 8 weeks ( in two treatment periods of four weeks, respectively) where patients will either maintain the previous dosage regimen or will step up to 20 mg per dose of vardenafil or will step down to 5 mg per dose of vardenafil, at interval visits of four weeks .

SUMMARY:
The primary objective of this study is to assess the efficacy together with safety of a flexible regimen, for a period of twelve weeks, of three doses (5 mg, 10mg and 20mg) of Bay 38-9456, a phosphodiesterase type V inhibitor, in males with erectile dysfunction treated with sildenafil in the previous <6 months .At entry, once the Inclusion and Exclusion criteria are confirmed, the study medication will be administered for twelve weeks in an open label design. Vardenafil will be administered, as needed, at a fix dose of 10 mg once daily for the first four weeks of treatment. At the Investigators' discretion, on the basis of efficacy and safety evaluations, the patients may, then, receive the same dose strength of their assigned study medication or, at the subsequent clinic visit(s), the next lower dose (5 mg vardenafil) or the next higher dose (20 mg vardenafil) for the subsequent four weeks of treatment. Previous dose level of vardenafil is either maintained, increased or decreased by one step according to the three applicable dose strengths (5 mg, 10 mg, 20 mg ). The highest dosage of vardenafil (20 mg) per day will not be exceeded. After twelve weeks of treatment, the patient will be contacted twenty four hours following the last visit in order to collect data concerning serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Males with erectile dysfunction for more than 6 months and no more than three years according to the NIH Consensus definition (the inability to achieve and maintain penile erection sufficient for satisfactory sexual intercourse)
* Stable, heterosexual relationship for more than 6 months
* Age range: 18 years and older
* Documented, written Informed Consent.

Exclusion Criteria:

A) Previous or current Medical Conditions

* Any unstable medical or psychiatric condition or substance abuse disorder that, in the opinion of the Investigator, is likely to affect the patient's ability to complete the study or precludes the patient's participation in the study
* Presence of penile anatomical abnormalities (e.g. penile fibrosis or Peyronie disease) that would significantly impair erectile function.
* Primary hypoactive sexual desire
* Erectile dysfunction after spinal cord injury
* Retinitis pigmentosa.
* History of positive test for Hepatitis B surface antigen (HbsAg) or Hepatitis C.
* Unstable angina pectoris
* History of myocardial infarction, stroke, electrocardiographic ischaemia (except stable angina), or life-threatening arrhythmia, within the prior 6 months.
* Atrial tachyarrhythmia (e.g. atrial fibrillation/flutter) with a heart rate of > 100 beats per minute at screening
* Severe chronic liver disease or liver function abnormalities
* Clinically significant chronic haematological disease or bleeding disorder
* History of significant peptic ulcer disease within one year of Visit 1.
* Resting hypotension (a resting systolic blood pressure of <90 mm Hg) or hypertension (a resting systolic blood pressure >170 mm Hg or a resting diastolic blood pressure >110 mm Hg)
* Symptomatic postural hypotension within the six months of Visit 1.
* Uncontrolled diabetes mellitus (Haemoglobin A1c > 12%)
* History of malignancy within the past 5 years (other than squamous or basal cell skin cancer and K prostatic).

B) Concomitant Medication 1. Patients who are taking nitrates or nitric oxide donors (e.g. molsidomine) .2. Patients who are taking anticoagulants, with the exception of anti-platelet agents.

3. Patients who are taking androgens (e.g. testosterone), trazodone or anti-androgens.

4. Patients who are taking the following potent inhibitors of cytochrome P 450 3A4: the HIV protease inhibitors ritonavir and indinavir, or the anti-mycotic agents itraconazole and ketoconazole (topical forms are allowed).

5. Patients who have received any investigational drug (including placebo) within 30 days of Visit 1.

6. Use of vardenafil (BAY 38-9456) at any time prior to the study. C) Abnormal Laboratory Values

1. Patients who have a serum total testosterone level >10% below the lower limit of normal (according to the range specified by the responsible laboratory).

2. Patients with serum creatinine > 2.5 mg/dL.D) Other Exclusion Criteria

1. Patients unwilling to cease use of vacuum devices, intracavernosal injection, Viagra or other therapy for erectile dysfunction for the entire course of the study .
2. Known hypersensitivity to any component of the investigational medication
3. Patients who are illiterate or are unable to understand the language in which the questionnaires are available.
4. Patients unwilling or unable to complete the patient diary card.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 527 (Actual)
Dates: Start 2003-05; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Percentage of success rate at the end of treatment period versus baseline. | At baseline, after 12 weeks

SECONDARY OUTCOMES:
The Erectile Function (EF) domain score of the International Index of Erectile Function (IIEF-Appendix 10.3) calculated as the sum of scores from Questions 1-5 and 15 at Visit 5 using the last Visit vs baseline. | Baseline, after 4 weeks, after 12 weeks
Global Assessment Question | Baseline, after 4 weeks, after 12 weeks
Italian validated Version of SF-12 Health Survey | Baseline, after 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer